CLINICAL TRIAL: NCT05817500
Title: Post-ICU Consultation : a Time to Discuss Advance Directives
Brief Title: Post-ICU Consultation : a Time to Discuss Advance Directives (CoPRADA)
Acronym: CoPRADA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0335 - CoPRADA
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Advance Directives; Post Intensive Care Syndrome; Advance Care Planning
Keywords: Intensive Care; Advance directives; Post Intensive Care syndrome; Post Intensive Care consultation
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients with > 48h mechanical ventilation and/or > 5 days stay in ICU

SUMMARY:
The aim of this study is to assess the possibility of discussing advance directives during post-intensive care consultation.

DETAILED DESCRIPTION:
After a stay in intensive care units (ICU), patients can experience physical, psychological and cognitive impairments. To assess this post intensive care syndrom (PICS), post-ICU consultation have been developed.

Since 5 year mortality is higher in ICU survivors, it might be interesting to address those patients' views relating to illness and end of life through a discussion on advance directives (AD), during post-ICU consultation.

However, the development of these consultations being recent, it has not yet been assessed whether this consultations might be a suitable time to discuss AD and the intensivit a suitable interlocutor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 48 hours of mechanical ventilation
* Patients with a 5 days stay in ICU

Exclusion Criteria:

* Patients with therapeutic limitation discussed during their ICU stay
* Geographical remotness to come to the post-ICU consultation
* Minor patients
* Patient not affiliated to the social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with at least 48 hours of mechanical ventilation and/or a 5 days stay in ICU, and then summoned to post-ICU consultation
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Number of patients willing to discuss AD after an ICU stay | 1 year
  Number of patient willing to discussion AD after ICU stay will be observed

SECONDARY OUTCOMES:
Number of patients knowing about AD before their ICU stay | 1 year
  Number of patient knowing before AD before ICU stay will be observed
Factors influencing the writing of AD after an ICU stay | 1 year
  Factors such as lenght of stay in ICU, lenght of hospitalisation, duration of mechanical ventilation /sedation and the existence of PTSD (PCLS) or anxiety/ depression (HADS) will be evaluated and their influence on the completion of AD
Evaluation of the privileged interlocutor to discuss AD | 1 year
  The privileged interlocutor to discuss AD will be observed
Evaluation of the privileged interlocutor to complete AD | 1 year
  The privileged interlocutor to complete AD will be observed

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rousseau AF, Prescott HC, Brett SJ, Weiss B, Azoulay E, Creteur J, Latronico N, Hough CL, Weber-Carstens S, Vincent JL, Preiser JC. Long-term outcomes after critical illness: recent insights. Crit Care. 2021 Mar 17;25(1):108. doi: 10.1186/s13054-021-03535-3. PMID 33731201
- [Background] Andreu P, Dargent A, Large A, Meunier-Beillard N, Vinault S, Leiva-Rojas U, Ecarnot F, Prin S, Charles PE, Fournel I, Rigaud JP, Quenot JP. Impact of a stay in the intensive care unit on the preparation of Advance Directives: Descriptive, exploratory, qualitative study. Anaesth Crit Care Pain Med. 2018 Apr;37(2):113-119. doi: 10.1016/j.accpm.2017.05.007. Epub 2017 Aug 4. PMID 28826983
- [Background] Lone NI, Walsh TS. Impact of intensive care unit organ failures on mortality during the five years after a critical illness. Am J Respir Crit Care Med. 2012 Oct 1;186(7):640-7. doi: 10.1164/rccm.201201-0059OC. Epub 2012 Jul 26. PMID 22837381